CLINICAL TRIAL: NCT01379144
Title: A 4 Week, Dose-Ranging, Multi-Center, Randomized, Double-Masked, Parallel Study Comparing The Efficacy, Safety, And Tolerability Of Latanoprost 75, 100 And 125 ug/ml To Xalatan In The Treatment Of Primary Open-Angle Glaucoma Aand Ocular Hypertension
Brief Title: A Study Comparing The Efficacy, Safety And Tolerability Of Latanoprost 75, 100 And 125 ug/ml To Xalatan In The Treatment Of Primary Open-Angle Glaucoma And Ocular Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XALA-0091-166; A6111066
Record Dates: First submitted 2011-06-20; First posted 2011-06-23 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2018-09

CONDITIONS: Primary Open Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Latanoprost

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- latanoprost 75 ug (Experimental)
  Interventions: Drug: latanoprost 75 ug
- latanoprost 100 ug (Experimental)
  Interventions: Drug: latanoprost 100 ug
- latanoprost 125 ug (Experimental)
  Interventions: Drug: latanoprost 125 ug
- latanoprost 50 ug (Active Comparator)
  Interventions: Drug: latanoprost 50 ug

INTERVENTIONS:
Drug: latanoprost 75 ug — Eligible patients were randomized to receive 1 of 4 different doses of latanoprost (50, 75, 100 or 125 ug/mL).
  Study medication was supplied in clear bottles. Patients were instructed to instill one drop of study medication in one or both eyes (as instructed by their investigator) once daily in the evening between 7 PM and 9 PM during the entire treatment period. The first dose of study medication was instilled in the evening of the baseline visit and the last dose was instilled in the evening before the Week 4 (Day 28) visit.
  Arms: latanoprost 75 ug
Drug: latanoprost 100 ug — Eligible patients were randomized to receive 1 of 4 different doses of latanoprost (50, 75, 100 or 125 ug/mL).
  Study medication was supplied in clear bottles. Patients were instructed to instill one drop of study medication in one or both eyes (as instructed by their investigator) once daily in the evening between 7 PM and 9 PM during the entire treatment period. The first dose of study medication was instilled in the evening of the baseline visit and the last dose was instilled in the evening before the Week 4 (Day 28) visit.
  Arms: latanoprost 100 ug
Drug: latanoprost 125 ug — Eligible patients were randomized to receive 1 of 4 different doses of latanoprost (50, 75, 100 or 125 ug/mL).
  Study medication was supplied in clear bottles. Patients were instructed to instill one drop of study medication in one or both eyes (as instructed by their investigator) once daily in the evening between 7 PM and 9 PM during the entire treatment period. The first dose of study medication was instilled in the evening of the baseline visit and the last dose was instilled in the evening before the Week 4 (Day 28) visit.
  Arms: latanoprost 125 ug
Drug: latanoprost 50 ug — Eligible patients were randomized to receive 1 of 4 different doses of latanoprost (50, 75, 100 or 125 ug/mL).
  Study medication was supplied in clear bottles. Patients were instructed to instill one drop of study medication in one or both eyes (as instructed by their investigator) once daily in the evening between 7 PM and 9 PM during the entire treatment period. The first dose of study medication was instilled in the evening of the baseline visit and the last dose was instilled in the evening before the Week 4 (Day 28) visit.
  Arms: latanoprost 50 ug

SUMMARY:
The primary objective of this study was to compare the change in intraocular pressure (IOP) of three different doses of latanoprost (75, 100 and 125 ug/ml) to that of the marketed 50 ug/ml dose, in a dose ranging study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older.
* Primary open angle glaucoma (POAG) or ocular hypertension (OHT) requiring unilateral or bilateral administration of intraocular pressure (IOP) lowering treatment, including patients who were naïve to IOP lowering treatment.
* IOP between ≥ 24 mmHg and ≤ 36 mmHg in at least one eye at the 8 AM time point at baseline/randomization.

Exclusion Criteria:

* Closed/barely open anterior chamber angle or a history of acute angle closure.
* A history of discontinued prostaglandin IOP lowering treatment, unless the reason for discontinuation was participation in a clinical study.
* Ocular surgery or argon laser trabeculoplasty in one or both eyes within 3 months prior to the screening visit.
* Use or anticipated requirement during the study of any topical medication that was known to affect IOP.
* Anticipated need to modify systemic medication known to affect IOP (eg, beta-adrenergic antagonists, alpha-adrenergic agonists, calcium channel blockers, angiotension converting enzyme inhibitors, and angiotension II receptor antagonists) during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2003-01; Primary Completion 2003-03 (Actual); Study Completion 2003-04 (Actual)

PRIMARY OUTCOMES:
The primary endpoint was the change in intraocular pressure (IOP) at 8 AM and 4 PM from baseline to Week 4 (Day 28). | Baseline and Day 28

SECONDARY OUTCOMES:
The change in intraocular pressure (IOP) at 8 AM and 4 PM from baseline across all clinic visits; comparisons were made by separate analyses for each time point and visit. | Baseline and Day 28
The percentage change in IOP from baseline at 8 AM to Week 4 (Day 28). | Baseline and Day 28
Ocular safety assessments (ie, ocular adverse events, assessment of conjunctival hyperemia, and ocular symptom evaluations) across all clinic visits. | Baseline and Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (25):
- Australia (3):
  - Eye Associates Pty Limited, Sydney, New South Wales
  - Save Sight Institute, Sydney, New South Wales
  - Royal Adelaide Hospital, North Terrace, Adelaide, South Australia
- Czechia (5):
  - University Hospital Brno-Bohunice, Brno
  - Specializovana Glaukomova Poradna, Blanicka 25, Prague
  - VseobecnBfakultnf nemocnice, Prague
  - Private Ophthalmology, V Hurkach 1296, Prague
  - Institute of Aviation Medicine, Generalal Piky 1, Prague
- France (4):
  - Hopital De La Timone, Marseille
  - Hopital Des Armees Laveran, Marseille
  - Fondation Adolphe De Rothchild, Paris
  - Hopital Civil, Strasbourg
- Akadimos Ophthalmology Center of Northern Greece, Thessaloniki, Greece
- Pakistan (4):
  - Layton Rahmatullah Benevolent Trust (LRBT), Eye Hospital, Lahore, Punjab Province
  - Services Hospital Lahore, Lahore, Punjab Province
  - Aga Khan University Hospital Karachi, Karachi, Sindh
  - Civil Hospital Karachi, Karachi, Sindh
- Portugal (3):
  - A.I.B.I.L.I., Coimbra
  - Hospital De S. Jose, Lisbon
  - Hospital Pedro Hispano, Matosinhos Municipality
- Thailand (2):
  - Siriraj Hospital, Ophthalmology, Bangkok
  - Chulalongkorn Hospital, Bangkok
- United Kingdom (3):
  - Birmingham Heartlands Hospital, Birmingham
  - Glasgow Royal Infirmary, Glasgow
  - Sunderland Eye Infirmary, Sunderland

REFERENCES:
- [Derived] Eveleth D, Starita C, Tressler C. A 4-week, dose-ranging study comparing the efficacy, safety and tolerability of latanoprost 75, 100 and 125 mug/mL to latanoprost 50 mug/mL (xalatan) in the treatment of primary open-angle glaucoma and ocular hypertension. BMC Ophthalmol. 2012 May 18;12:9. doi: 10.1186/1471-2415-12-9. PMID 22607109
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=XALA-0091-166